CLINICAL TRIAL: NCT03348228
Title: Effect of Hydroxycitrate on Urine Chemistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00147
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Nephrolithiasis
Keywords: Hydroxycitrate Supplements
MeSH Terms: conditions — Nephrolithiasis | interventions — hydroxycitric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Participants willrecord a self-selected diet for 3 days and then perform two 24-hour urine collections on the last 2 days of this diet. HCA will be administered afterwards to both groups (see methods below) for 7 days
  Interventions: Dietary Supplement: Hydroxycitrate (HCA)
- Calcium Stone Formers (Active Comparator): Participants willrecord a self-selected diet for 3 days and then perform two 24-hour urine collections on the last 2 days of this diet. HCA will be administered afterwards to both groups (see methods below) for 7 days
  Interventions: Dietary Supplement: Hydroxycitrate (HCA)

INTERVENTIONS:
Dietary Supplement: Hydroxycitrate (HCA) — Hydroxycitrate supplements are available over the counter and are primarily promoted as a weight loss supplement. Each subject will be given 42 capsules of Swanson super citrimax (hydroxycitrate) Details of the product are provided above. The subjects will be asked to take the capsules over a seven period (6 capsules per day).

SUMMARY:
Hydroxycitrate (HCA) is a compound extracted from the fruit, Garcinia Cambogia. Hydroxycitrate supplements are available over the counter and are primarily promoted as a weight loss supplement. There has been recent evidence that hydroxycitrate is a potent inhibitor of calcium oxalate crystal growth and can lead to the dissolution of the crystals. The purpose of this research study is to study the effect of Hydroxycitrate (HCA) supplements on HCA urinary excretion and on urine chemistries in kidney stone formers and normal subjects.

ELIGIBILITY:
Inclusion Criteria:

Stone formers group:

* Established diagnosis of recurrent calcium stone formers
* Ages between 18 and 80
* Subjects must be able to read and follow instructions clearly and able to do 24 hour urine collections.
* Subjects must be voluntarily willing and able to sign an informed consent form.

Control Group:

* In addition to b, c and d above, subjects must not have any known kidney disease or family history of renal stones. Inclusion would be based on information provided by participants.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
changes in urinary excretion of citrate | 7 Days
  Paired t-tests will be performed to compare any changes in citrate before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: David Goldfarb, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided